CLINICAL TRIAL: NCT00276757
Title: Treatment Protocol of the Third International Study For Langerhans Cell Histiocytosis
Brief Title: Combination Chemotherapy in Treating Young Patients With Langerhans Cell Histiocytosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Histiocyte Society (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000454768; HISTSOC-LCH-III; CCLG-LCH-III; EU-20587; CCLG-LCH-2002-07; UMN-2006NT004
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2007-05

CONDITIONS: Childhood Langerhans Cell Histiocytosis
Keywords: childhood Langerhans cell histiocytosis
MeSH Terms: interventions — Leucovorin; Methotrexate; Prednisolone; Vinblastine

INTERVENTIONS:
Drug: leucovorin calcium
Drug: methotrexate
Drug: prednisolone
Drug: vinblastine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of Langerhans cell histiocytosis, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may be an effective treatment for Langerhans cell histiocytosis.

PURPOSE: This randomized clinical trial is studying combination chemotherapy to see how well it works in treating young patients with Langerhans cell histiocytosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy, in terms of response to initial therapy, of prednisolone, vinblastine, and mercaptopurine with vs without methotrexate and leucovorin calcium in young patients with Langerhans cell histiocytosis.
* Compare the progression-free survival of patients with low-risk Langerhans cell histiocytosis who responded to initial therapy who are then treated with 6-month vs 12-month continuation therapy comprising prednisolone and vinblastine.

Secondary

* Compare the acute and long-term toxicity and the incidence of permanent effects.
* Compare the overall and progression-free survival, response rate, and time until response.

OUTLINE: This is a randomized, multicenter study with one pilot nonrandomized stratum. Patients are stratified according to number of systems involved (multiple vs single) and organs involved (at risk vs low risk).

* Stratum 1 (at risk patients): Patients are further stratified according to participating center. Patients are randomized to 1 of 2 treatment arms (arms I and II).

  * Arm I:

    * Initial therapy: Patients receive oral prednisolone 3 times daily on days 1-28 followed by a taper on days 29-42 and vinblastine IV on days 1, 8, 15, 22, 29, and 36. Patients achieving nonactive disease (NAD) after course 1 proceed to continuation therapy. Patients achieving intermediate response or disease regression receive a second course* of initial therapy. Patients achieving NAD or disease regression after course 2 proceed to continuation therapy.
    * Continuation therapy: Patients receive oral mercaptopurine daily for 3 weeks, pulsed oral prednisolone 3 times daily on days 1-5, and vinblastine IV on day 1. Treatment repeats every 3 weeks until day 365 from the beginning of therapy in the absence of disease progression or unacceptable toxicity.
  * Arm II:

    * Initial therapy: Patients receive prednisone and vinblastine as in arm I initial therapy. Patients also receive methotrexate IV over 24 hours on days 1, 15, and 29 and oral leucovorin calcium twice daily on days 2,16, and 30. Patients achieving NAD after course 1 proceed to continuation therapy. Patients achieving intermediate response or disease regression receive a second course* of initial therapy. Patients achieving NAD or disease regression after course 2 proceed to continuation therapy.
    * Continuation therapy: Patients receive oral mercaptopurine daily for 3 weeks, pulsed oral prednisolone 3 times daily on days 1-5, vinblastine IV on day 1, and oral methotrexate on day 1. Treatment repeats every 3 weeks until day 365 from the beginning of therapy in the absence of disease progression or unacceptable toxicity.
* Stratum 2 (low-risk patients): Patients are stratified according to age at diagnosis (≤ 2 vs > 2) and participating center. Patients are randomized to 1 of 2 treatment arms (arms III and IV) after the first course of initial therapy.

  * Arm III:

    * Initial therapy: Patients receive prednisolone and vinblastine as in course 1 of stratum 1 arm I initial therapy. Patients achieving NAD or disease regression after course 1 proceed to continuation therapy. Patients achieving intermediate or worse response receive a second course* of initial therapy. Patients achieving NAD, disease regression, or intermediate response after course 2 proceed to continuation therapy.
    * Continuation therapy: Patients receive prednisolone and vinblastine as in stratum 1 arm I continuation therapy. Treatment continues until day 182 from the beginning of initial therapy in the absence of disease progression or unacceptable toxicity.
  * Arm IV:

    * Initial therapy: Patients receive 1-2 courses of prednisolone and vinblastine as in stratum 2 arm III.
    * Continuation therapy: Patients receive pulsed prednisolone and vinblastine as in stratum 1 arm I continuation therapy. Treatment continues until day 365 from the beginning of initial therapy in the absence of disease progression or unacceptable toxicity.
* Stratum 3 (pilot study) (patients with multifocal bone disease and/or special sites):

  * Initial therapy: Patients receive prednisolone and vinblastine as in stratum 1 arm I initial therapy. Patients achieving NAD or disease regression after course 1 proceed to continuation therapy. Patients with disease progression receive a second course* of initial therapy. Patients achieving NAD or disease regression after course 2 proceed to continuation therapy.
  * Continuation therapy: Patients receive pulsed prednisolone and vinblastine as in stratum 1 arm I continuation therapy. Treatment continues until day 182 from the beginning of initial therapy in the absence of disease progression or unacceptable disease.

NOTE: *Patients receive oral prednisolone 3 times daily on days 43-45, 50-52, 57-59, 64-66, 71-73, and 78-80 only during the second course of initial therapy.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 376 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histopathologically confirmed diagnosis of Langerhans cell histiocytosis according to the criteria defined by the Histiocyte Society

  * Demonstration of CD1a antigenic determinants on the surface of lesional cells (by immunocytology or immunohistology) or Birbeck granules in lesional cells by electron microscopy
* Considered at risk or low risk according to the following criteria:

  * Multi-system at risk disease, defined as involvement of one or more risk organs (i.e., hematopoietic system, liver, spleen, or lungs)

    * No single-system lung involvement
  * Multi-system low-risk disease

    * Multiple organs involved but without involvement of risk organs
  * Single-system disease

    * Multifocal bone disease (i.e., lesions in 2 or more different bones)
    * Localized special site involvement, such as CNS-risk lesions with intracranial soft tissue extension or vertebral lesions with intraspinal soft tissue extension

      * Vault lesions are not regarded as CNS-risk lesions

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior treatment for Langerhans cell histiocytosis

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 376 (Estimated)
Dates: Start 2001-04; Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L. McClain, MD, PhD, Study Chair — Texas Children's Cancer Center
Locations (33):
- United States (4):
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas
- Hospital de Pediatria Garrahan, Buenos Aires, Buenos Aires, Argentina
- St. Anna Children's Hospital, Vienna, Austria
- Hospital for Sick Children, Toronto, Ontario, Canada
- CHR Hotel Dieu, Nantes, France
- University Medical Center Hamburg - Eppendorf, Hamburg, Germany
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia, Italy
- Karolinska University Hospital - Solna, Stockholm, Sweden
- United Kingdom (21):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Children's Cancer and Leukaemia Group, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales

REFERENCES:
- [Derived] Gadner H, Minkov M, Grois N, Potschger U, Thiem E, Arico M, Astigarraga I, Braier J, Donadieu J, Henter JI, Janka-Schaub G, McClain KL, Weitzman S, Windebank K, Ladisch S; Histiocyte Society. Therapy prolongation improves outcome in multisystem Langerhans cell histiocytosis. Blood. 2013 Jun 20;121(25):5006-14. doi: 10.1182/blood-2012-09-455774. Epub 2013 Apr 15. PMID 23589673